CLINICAL TRIAL: NCT03016052
Title: Visual Mismatch Negativity in Attention Bias Modifcation Treatment for Social and Generalized Anxiety- an ERP Study
Brief Title: Visual Mismatch Negativity in Attention Bias Modifcation Treatment for Anxiety
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tel Aviv University (Other)
Responsible Party: Principal Investigator, Yair Bar-Haim, Professor, Tel Aviv University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TAUvMMN
Record Dates: First submitted 2017-01-08; First posted 2017-01-10 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-11

CONDITIONS: Social Anxiety Disorder; Generalized Anxiety Disorder
Keywords: ABMT; social anxiety; generalized anxiety
MeSH Terms: conditions — Phobia, Social; Generalized Anxiety Disorder

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ABMT (Experimental): The attention bias modification treatment comprises of six computerized sessions, twice a week, in purpose of modulate biases in attention for threat stimuli.
  Interventions: Behavioral: ABMT

INTERVENTIONS:
Behavioral: ABMT — Participants will be trained with a dot-probe task including angry-neutral faces. The task will be adapted for the oddball paradigm, such that in 80% of trials the probe will appear in place of the neutral face, and in 20% of trials in place of the angry face.
  Other Names: attention bias modification

SUMMARY:
this study examines the emergence of the visual mismatch negativity (vMMN) ERP component in response to deviations from the embedded contingency in attention bias modification treatment (ABMT) for social and generalized anxiety, and the interaction between vMMN emergence and clinical improvement.

***As of September 2017, recruitment of SAD participants has concluded.

DETAILED DESCRIPTION:
all participants, suffering from either social anxiety disorder or generalized anxiety disorder, will receive 6 sessions of ABMT, adapted for an oddball paradigm. two of the sessions will also include simultaneous EEG measurement. the goal of the study is to determine the emergence of vMMN in response to trials deviating the embedded contingency and to examine the correlation between vMMN emergence and clinical improvement of anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

* A signed consent form
* Men and women between the ages of 18 and 65.
* Meeting a current diagnosis of Social Anxiety Disorder (SP) or Generalized Anxiety Disorder according to the DSM-IV
* SP/GAD as the primary diagnosis: In cases of co-morbidity, SP/GAD will be deemed as the most distressing and clinically significant condition among the co-morbid disorders.
* Stable pharmaco-therapy: Participants receiving a pharmacological treatment who are taking a stable medication for at least 3 months before the beginning of the procedure.

Exclusion Criteria:

* A diagnosis of psychotic or bipolar disorders.
* A diagnosis of a neurological disorder (i.e., epilepsy, brain injury).
* Drug or alcohol abuse.
* A pharmacological treatment that is not stabilized in the past 3 months.
* Another psychotherapeutic treatment.
* Change in treatment during the study.
* Poor judgment capacity (i.e., children under 18 and special populations).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
Change from baseline - the Liebowitz Social Anxiety Scale - Diagnostic Interview scores | 1 week after treatment completion and 2 months after treatment completion
  The LSAS is a 24-item scale, each item corresponding to a situation selected on the basis of clinical experience. Each item is rated on a severity scale ranging from 0 to 3 with regard to the passing week, measuring separately two components of social anxiety, specifically, fear/anxiety and avoidance of social interaction and performance situations. Although the assessor may request and ask for further detail and adjust the rating based on clinical experience, this option is not often exercised, and inter-rater agreement is not considered to be a relevant concern.
Change from baseline - The Generalized Anxiety Disorder Severity Scale | 1 week after treatment completion and 2 months after treatment completion
  The Generalized Anxiety Disorder Severity Scale (GADSS) is a 6-item interview assessment that evaluates the severity of each of the DSM-IV symptoms of generalized anxiety disorder. It begins with a target worry list to identify situations that are the focus of worry, and continues with six 5-point-scale items to evaluate levels of generalized anxiety severity.

SECONDARY OUTCOMES:
Change from baseline - the Social Phobia Inventory scores | 1 week after treatment completion and 2 months after treatment completion
  This is a 17-item self-report measure of social anxiety evaluating fear, avoidance and physiological discomfort. Each item is rated on scale ranging from 0 to 4 with a possible total score of 68.
Change from baseline - the Penn State Worry Questionnaire | 1 week after treatment completion and 2 months after treatment completion
  This is a 16-item self-report measure of the worry dimension of generalized anxiety disorder. the questionnaire is composed of statements, and subjects are request to rate how typical each item is of them, ona 5-point scale ranging from "not typical at all" to "very typical". the PSWQ includes 5 reverse questions.
Change from baseline - the GAD-7 | 1 week after treatment completion and 2 months after treatment completion
  This is a 7-item self-report measure of generalized anxiety. Each item is rated on a 4-point scale with a possible score of 0-21. Increasing scores indicating increased functional impairment.

OTHER OUTCOMES:
changes in the Mini-International Neuropsychiatric Interview (M.I.N.I) diagnosis | 1 week after treatment completion and 2 months after treatment completion
  structured diagnostic interview for DSM - IV and ICD-10 psychiatric disorders, which takes approximately 20 min to administer and is a valid and time-efficient alternative to the SCID-P and CIDI.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Bar-Haim, PhD, Principal Investigator — Tel Aviv University
Locations (1):
- Tel Aviv University, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No